CLINICAL TRIAL: NCT07116941
Title: Effects of Multisensory and Cognitive Interventions Applied in the Intensive Care Unit on Physiological, Psychological and Functional Outcomes
Brief Title: Multisensory and Cognitive Interventions in the ICU: Effects on Health and Recovery
Acronym: MICU-CARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Alp Ozel, Assistant Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AIBU-FTR-AO-04
Record Dates: First submitted 2025-07-25; First posted 2025-08-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Coronary Artery Bypass Graft (CABG); Cardiac Surgery Subjects; Postoperative Care
Keywords: Early Mobilization; Intensive Care Unit; Cardiac Surgery; Multisensory Intervention; Anxiety; Non-pharmacological Intervention; Rehabilitation in ICU
MeSH Terms: conditions — Anxiety Disorders | interventions — Acoustic Stimulation

STUDY DESIGN:
Intervention Model Description: This study is a prospective, randomized, controlled, parallel-group clinical trial with four arms. Participants are randomly assigned to one of the following groups: control (standard ICU care), cognitive stimulation, auditory stimulation, or multisensory stimulation. Each participant receives a single type of intervention without crossover. Interventions are delivered during the early mobilization (sitting) phase in the ICU. Randomization is performed using a computer-generated allocation sequence, and outcome assessors are blinded to group assignments.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors are blinded to group allocation. Interventions are administered by a separate team of staff members who are not involved in outcome assessment. Participants are unaware of the specific intervention purpose and content, and standard instructions are used across all groups to minimize expectancy bias. Care providers are not blinded due to the nature of the interventions, but contact with assessors is minimized to maintain blinding integrity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (No Intervention): Participants will receive standard ICU care without any additional cognitive or sensory stimulation during the sitting phase of early mobilization.
- Cognitive Stimulation Group (Experimental): Participants will perform simple cognitive exercises (e.g., word games, attention tasks, problem solving) during a 30-minute sitting session in the ICU.
  Interventions: Behavioral: Cognitive Exercises
- Auditory Stimulation Group (Experimental): Participants will listen to calming music or nature sounds via headphones for 30 minutes during the sitting phase in the ICU.
  Interventions: Behavioral: Auditory Stimulation
- Multisensory Stimulation Group (Experimental): Participants will receive tactile stimulation using hand therapy balls and olfactory stimulation using lavender or mint scent for 30 minutes during the sitting phase in the ICU.
  Interventions: Behavioral: Multisensory Stimulation

INTERVENTIONS:
Behavioral: Cognitive Exercises — Participants perform a 30-minute session of cognitive tasks during the sitting phase of early ICU mobilization. Activities include word games, attention exercises, and simple problem-solving tasks designed to engage memory and executive function.
  Arms: Cognitive Stimulation Group
Behavioral: Auditory Stimulation — Participants listen to calming music or nature sounds through headphones for 30 minutes during early mobilization in the ICU. The auditory content is selected to reduce anxiety and promote relaxation.
  Arms: Auditory Stimulation Group
Behavioral: Multisensory Stimulation — Participants receive 30 minutes of combined sensory stimulation during the sitting phase in the ICU. This includes tactile stimulation using hand therapy balls and olfactory stimulation with lavender or mint-scented materials to enhance relaxation and sensory engagement.
  Arms: Multisensory Stimulation Group

SUMMARY:
The goal of this clinical trial is to examine the effects of sensory and cognitive stimulation on physiological, psychological, and functional recovery in adult patients after cardiac surgery who are treated in the intensive care unit (ICU). The main questions it aims to answer are:

* Does sensory and/or cognitive stimulation reduce anxiety and improve hemodynamic stability in ICU patients?
* Does it enhance physical function and independence during early rehabilitation in the ICU?

Researchers will compare four groups:

1. Standard care (control),
2. Cognitive stimulation,
3. Auditory stimulation (music),
4. Multisensory stimulation (touch + smell)

to assess which intervention is most effective in improving recovery parameters.

Participants will:

* Be randomly assigned to one of four groups during early mobilization in the ICU
* Receive a 30-minute intervention session depending on group assignment
* Be evaluated for heart rate, blood pressure, oxygen saturation, anxiety (VAS), physical function (PFIT, FIM), and satisfaction before and after the session

DETAILED DESCRIPTION:
This randomized controlled trial aims to evaluate the effects of sensory and cognitive stimulation interventions on physiological, psychological, and functional recovery in adult patients who have undergone cardiac surgery and are admitted to the intensive care unit (ICU). Despite early mobilization protocols being widely adopted in ICU settings, the added value of non-pharmacological interventions such as auditory, tactile, olfactory, and cognitive stimulation has not been comprehensively studied in the context of intensive care recovery.

The study addresses the gap in clinical practice regarding multisensory deprivation in ICUs, which can lead to heightened anxiety, delayed functional recovery, and impaired hemodynamic regulation. Previous research has suggested that music therapy, aromatherapy, tactile stimulation, and cognitive exercises may provide benefit individually. However, comparative or combined effects of these modalities remain unexplored in a structured clinical design.

Participants will be randomly assigned to one of four groups: control (standard ICU care), cognitive stimulation, auditory stimulation (music or nature sounds), and multisensory stimulation (lavender or mint aroma combined with tactile stimulation using hand therapy balls). Each intervention will be administered for 30 minutes during the sitting phase of early mobilization.

The primary outcome is improvement in functional independence measured by the Functional Independence Measure (FIM). Secondary outcomes include physiological parameters (heart rate, blood pressure, oxygen saturation, respiratory rate), psychological outcomes (anxiety level assessed by VAS, patient satisfaction), and functional capacity (ICU sitting tolerance, PFIT scores). Assessments will be conducted before, immediately after, and 15 minutes following the intervention to capture both immediate and delayed effects.

The findings of this study are expected to contribute to evidence-based rehabilitation strategies in critical care settings and offer low-cost, non-invasive interventions that can be easily integrated into standard ICU practice to enhance patient comfort and recovery.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* Underwent coronary artery bypass grafting (CABG) or other open-heart surgery
* Admitted to the ICU postoperatively and eligible for early mobilization
* Hemodynamically stable (within normal blood pressure and heart rate ranges, without inotropic support)
* Alert and able to communicate

Exclusion Criteria:

* Diagnosis of ICU delirium or altered mental status
* Severe hemodynamic instability
* Presence of neurological disease or significant cognitive impairment
* Significant sensory deficits (e.g., severe hearing or vision loss)
* Known allergy or psychological sensitivity to auditory or olfactory stimuli (e.g., aromatherapy or music)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Functional Independence Measure (FIM) Total Score | Change in outcome measures from baseline (24 hours post-surgery, prior to intervention), to immediately after intervention (within 1 minute), and at hospital discharge (approximately postoperative Day 5-7).
  Functional recovery will be assessed using the Functional Independence Measure (FIM), which comprises 18 items evaluating motor and cognitive functions. Each item is scored on a 7-point scale, yielding a total score ranging from 18 (complete dependence) to 126 (complete independence), with higher scores indicating greater independence.

SECONDARY OUTCOMES:
Visual Analog Scale for Anxiety Assessment | Change in outcome measures from baseline (24 hours post-surgery, prior to intervention), to immediately after intervention (within 1 minute), and 15 minutes after intervention
  Anxiety will be assessed using the Visual Analog Scale (VAS), which consists of a 10-centimeter horizontal line anchored with "no anxiety" (score = 0) on the left end and "worst imaginable anxiety" (score = 10) on the right end. Patients will be instructed to place a mark on the line that best represents the intensity of their current anxiety. The score will be determined by measuring the distance in centimeters from the left end of the line to the point marked by the patient. Higher scores indicate greater levels of anxiety.
Heart Rate | Heart rate will be recorded at three time points: before the intervention, immediately after the session, and 15 minutes post-intervention.
  Heart rate (beats per minute, bpm) will be measured to assess the autonomic physiological response to the intervention. Measurements will be performed using a standard bedside patient monitor while the participant is in a seated resting position. Changes in heart rate may reflect autonomic activation or relaxation in response to the intervention.
Blood Pressure | Blood pressure will be recorded at three time points: before the intervention, immediately after the session, and 15 minutes post-intervention.
  Blood pressure (systolic and diastolic, mmHg) will be measured to evaluate the cardiovascular response to the intervention. Measurements will be obtained using a calibrated automatic sphygmomanometer while the participant is in a seated resting position, with the arm supported at heart level. Variations in systolic and/or diastolic values may indicate hemodynamic responses related to stress or relaxation.
Respiratory Rate | Respiratory rate will be recorded at three time points: before the intervention, immediately after the session, and 15 minutes post-intervention.
  Respiratory rate (breaths per minute) will be measured to assess the respiratory response to the intervention. Measurements will be performed using a standard bedside patient monitor while the participant is in a seated resting position. An increase or decrease in respiratory rate may reflect physiological arousal or relaxation in response to the intervention.
Oxygen Saturation | SpO₂ values will be recorded at three time points: before the intervention, immediately after the session, and 15 minutes post-intervention.
  Oxygen saturation (SpO₂, %) will be measured to assess peripheral oxygenation status in response to the intervention. Measurements will be obtained using a standard pulse oximeter while the participant is in a seated resting position. igher values indicate better oxygenation, while decreases may reflect impaired respiratory function or increased physiological demand. A change greater than 4 percentage points will be considered clinically significant.
Patient Satisfaction Score | Immediately after and 15 minutes after intervention
  Satisfaction will be assessed using a 5-item questionnaire, with each item rated from 1 (strongly disagree) to 5 (strongly agree). The mean score will be calculated.
Physical Function in Intensive Care Test | Change in outcome measures from baseline (24 hours post-surgery, prior to intervention) to immediately after intervention (within 1 minute)
  The Physical Function in Intensive Care Test (PFIT) is a performance-based measure used to assess physical function in critically ill patients. It evaluates four components: sit-to-stand assistance, marching on the spot (cadence), shoulder (or quadriceps) strength, and duration of marching. Each component is scored and combined into a total PFIT score ranging from 0 to 12. Higher scores indicate better physical function and greater mobility capacity.
Sitting Tolerance Time | During the intervention session
  Duration (in minutes and seconds) that participants can maintain a seated position will be recorded. Criteria include hemodynamic stability and subjective tolerance (e.g., dizziness, fatigue).

CONTACTS AND LOCATIONS:
Overall Officials: Alp Ozel, PT, PhD, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Bolu Abant Izzet Baysal University, Izzet Baysal Training and Research Hospital, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in this study will be shared after de-identification. The data will be made publicly available at the time of publication via the Zenodo online repository (https://zenodo.org).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: IPD and supporting documents will be available starting at the time of publication and will remain indefinitely accessible via the Zenodo repository (https://zenodo.org).
Access Criteria: The individual participant data (IPD) and supporting documents (including the study protocol, statistical analysis plan, and analytic code) will be publicly accessible to anyone via the Zenodo repository (https://zenodo.org) without restriction.
URL: https://zenodo.org/